CLINICAL TRIAL: NCT01321827
Title: Monotherapy of Itraconazole Versus Prednisolone in Allergic Bronchopulmonary Aspergillosis
Acronym: MIPA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IGCST; MS/1398/Res/1838 (Other: PGIMER)
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Allergic Bronchopulmonary Aspergillosis
Keywords: ABPA
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary | interventions — Glucocorticoids; Prednisolone; Itraconazole; Azoles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Itraconazole group (Experimental): Itraconazole 200 mg BD for 4 months along with inhaled formoterol/fluticasone (6/125 mcg) 2 puffs twice daily by MDI and as needed as per the SMART approach
  Interventions: Drug: Itraconazole
- Glucocorticoid group (Active Comparator): Prednisolone 0.5 mg/kg/day for 4 weeks; 0.25 mg/kg/day for 4 weeks; 0.125 mg/kg/day for 4 weeks. Then taper by 5 mg every 2 weeks and discontinue. Patients will also receive inhaled formoterol/fluticasone (6/125 mcg) as needed as per the SMART approach for control of asthma
  Interventions: Drug: Glucocorticoids

INTERVENTIONS:
Drug: Glucocorticoids — Prednisolone 0.5 mg/kg/day for 4 weeks; 0.25 mg/kg/day for 4 weeks; 0.125 mg/kg/day for 4 weeks. Then taper by 5 mg every 2 weeks and discontinue. Patients will also receive inhaled formoterol/fluticasone (6/125 mcg) as needed as per the SMART approach for control of asthma
  Other Names: Prednisolone
  Arms: Glucocorticoid group
Drug: Itraconazole — Itraconazole 200 mg BD for 6 months along with inhaled formoterol/fluticasone (6/125 mcg) 2 puffs twice daily by MDI and as needed as per the SMART approach
  Other Names: Azole
  Arms: Itraconazole group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of itraconazole monotherapy in patients with ABPA.

DETAILED DESCRIPTION:
Allergic bronchopulmonary aspergillosis (ABPA) is a pulmonary disorder caused by a complex hypersensitivity response to antigens released by the fungus Aspergillus fumigatus. The clinical entity was first described by Hinson et al in 1952, and the clinical and immunologic significance of Aspergillus fumigatus in the sputum were reported by Pepys and coworkers in 1959. The prevalence of ABPA in bronchial asthma is fairly high and a recent meta-analysis suggested the prevalence of ABPA in asthma clinics to be as high as 13 percent. Diagnostic criteria for ABPA have been laid and generally include the following eight major criteria: (a) history of asthma; (b) transient or fixed pulmonary infiltrates; (c) immediate cutaneous hyperreactivity to A fumigatus antigen; (d) absolute eosinophil count > 1000/µL; (e) serum precipitins against A fumigatus; (f) total IgE levels > 1000 IU/mL; (g) central bronchiectasis on high-resolution computed tomography (HRCT); and, (h) raised A fumigatus specific IgE or IgG levels. However, none of these are specific for ABPA,and there is still no consensus on the number of criteria needed for diagnosis, and patients in different stages of ABPA may not fulfill all these criteria. Also, there is no established definition for remission of ABPA. The most widely followed criteria are clinical and radiological improvement with at least 35 percent decline in total serum IgE levels. However, in a recent study the investigators demonstrated that a 35% decline in serum IgE levels at six weeks is not seen in all patients with ABPA, and the decline is slower in patients with baseline IgE levels < 2500 IU/mL. Moreover, the quantum decline in serum IgE levels did not predict clinical outcome. The disorder is highly prevalent in India. The investigators have previously reported our experience with screening stable outpatients with bronchial asthma and acute severe asthma for ABPA. The investigators have also recently reported the prognostic factors associated with clinical outcomes in patients with ABPA.

Oral corticosteroids are currently the treatment of choice for ABPA associated with bronchial asthma. They not only suppress the immune hyperfunction but are also anti-inflammatory. However, there is no data to guide the dose and duration of glucocorticoids and different regimens of glucocorticoids have been used in literature. Itraconazole, an oral triazole with relatively low toxicity, is active against Aspergillus spp. in vitro and in vivo. The activity of itraconazole against Aspergillus spp. is more than that of ketoconazole. The administration of itraconazole can eliminate Aspergillus in the airways and can theoretically reduce the allergic responses in ABPA. The aim of this prospective randomized controlled trial (RCT) is to evaluate the efficacy and safety of itraconazole monotherapy in patients with ABPA.

ELIGIBILITY:
Inclusion Criteria: Patients will be included in the study if they meet the criteria for ABPA defined by

Presence of all the following three criteria:

* immediate cutaneous hyperreactivity on aspergillus skin test
* elevated total IgE levels > 1000 IU/mL
* A fumigatus specific IgE levels > 0.35 kU/L

Two of the following criteria:

* presence of serum precipitating antibodies against A fumigatus
* fixed or transient radiographic pulmonary opacities
* absolute eosinophil count > 1000/µL
* central bronchiectasis on HRCT.

Exclusion Criteria:

* if they have taken glucocorticoids for more than three weeks in the preceding six months
* failure to give informed consent
* enrollment in another trial of ABPA

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Remission rates in the two groups at six weeks and three months | 6 weeks, 3 months
  Remission - if the IgE levels decline by >=25% and there is clinical improvement with partial/total clearance of chest radiographic lesions after three months of glucocorticoids (if previously present pulmonary opacities)
Percentage decline in IgE levels at six weeks and three months | 6 weeks, 3 months
  IgE levels will be noted at baseline six weeks and three months after glucocorticoid therapy and percentage decline will be calculated as: (baseline IgE levels minus IgE levels after six weeks of treatment) divided by baseline IgE levels
Complete remission rates in the two groups | 3 months, 6 months
  No ABPA exacerbations over the next 3 months after stopping therapy

SECONDARY OUTCOMES:
Relapse rates in the two groups at six and 12 months after completion of treatment | 6 months, 12 months
  Relapse - doubling of the baseline IgE levels irrespective of the patient's symptoms or appearance of radiologic infiltrates
Treatment related adverse effects in the two groups | Every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ritesh Agarwal, MD, DM, Principal Investigator — PGIMER, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Uttarakhand, India

REFERENCES:
- [Derived] Agarwal R, Dhooria S, Singh Sehgal I, Aggarwal AN, Garg M, Saikia B, Behera D, Chakrabarti A. A Randomized Trial of Itraconazole vs Prednisolone in Acute-Stage Allergic Bronchopulmonary Aspergillosis Complicating Asthma. Chest. 2018 Mar;153(3):656-664. doi: 10.1016/j.chest.2018.01.005. Epub 2018 Jan 11. PMID 29331473